CLINICAL TRIAL: NCT04351542
Title: Ayurveda for Flu-like Illness During the Covid 19 Outbreak: Non Randomised Single-blind Controlled Trial
Brief Title: Ayurveda for Flu Like Illness During Covid-19 Outbreak
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarogyam UK (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AU09
Record Dates: First submitted 2020-04-14; First posted 2020-04-17 (Actual); Last update posted 2020-04-17 (Actual); Status verified 2020-04

CONDITIONS: Flu Like Illness
MeSH Terms: interventions — Medicine, Ayurvedic

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Ayurveda care provide was blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ayurveda Care Group (Experimental): Individualised ayurveda treatment was given to participants based on individual constitution.
  Interventions: Dietary Supplement: Ayurveda; Other: Usual Care
- Usual Care Group (Active Comparator): Participants followed the usual care.
  Interventions: Other: Usual Care

INTERVENTIONS:
Dietary Supplement: Ayurveda — Based on individual constitution (ayurveda based assessment) and symptoms an individual has, ayurveda herbal supplement and self managed practices were advised along with usual care recommendation.
  Arms: Ayurveda Care Group
Other: Usual Care — Usual care recommended by National Health Services, self isolation, plenty fluid, rest and Paracetamol. During the Covid 19 outbreak, additional recommendation were followed given by health services.

SUMMARY:
This study aimed to evaluate the efficacy and safety of Ayurveda in reducing symptoms of flu like illness during the Covid 19 outbreak.

ELIGIBILITY:
Inclusion Criteria:

* Patients with fu like symptoms within 48 hours of onset during March2020
* Mild to moderate symptoms who were advised to self isolate at home for 7-14 days
* Flu like symptoms present at least one respiratory symptom (e.g. cough, nasal obstruction, sore throat) and at least one constitutional symptom other than fever (e.g. fatigue, headache, myalgias) of less than 48-hour duration
* Willing to consent and follow up

Exclusion Criteria:

* Pregnant/lactating

  * Participants with chronic pulmonary diseases or critical condition or already developed severe respiratory distress
  * Clinically malignancies, systemic infection, other medical or psychiatric condition which places the subject at unacceptable risk to participate in the study - Known hypersensitivity to any ayurveda herbal substances
* Severe symptoms of respiratory distress patients deemed to require intensive care immediately

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-04-12 (Actual)

PRIMARY OUTCOMES:
Time to achieve afebrile | Change from baseline to 3rd and 7th-day
  Time to bring down a fever (oral temperature < 37.2 ̊C)
Severity of symptom score | Change from baseline to 3rd and 7th day
  Symptoms diary card completed twice daily from Day 0 to Day 7

SECONDARY OUTCOMES:
Patient reported improvement | Change from baseline to 3rd and 7th-day
  Patient reported improvement using 4 scale; 0-none, 1-weak, 2-medium, 3-strong

CONTACTS AND LOCATIONS:
Overall Officials: Neha Sharma, PhD, Principal Investigator — Aarogyam UK; Jaydeep Joshi, BAMS, Study Director — Aarogyam UK
Locations (1):
- Aarogyam, Leicester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided